CLINICAL TRIAL: NCT03569904
Title: Markers of Pulmonary Dysbiosis Associated With Exacerbation in Patients Followed for Cystic Fibrosis
Acronym: DYSBIOSE-CF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.317
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Cystic Fibrosis Pulmonary Exacerbation
Keywords: Cystic fibrosis; Pulmonary Dysbiosis; pulmonary exacerbation; Fungal bacterial pulmonary dysbiosis; Viral bacterial pulmonary dysbiosis; Microbiota
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim objective is to identify markers of bacterial, viral and fungal pulmonary dysbiosis, associated with the occurrence of exacerbation in patients followed for cystic fibrosis.

The primary endpoint is the association between a modification of at least 10% of the relative abundance of a bacterial phylum (Proteobacteria, Firmicutes, Actinobacteria, Bacteroidetes, Fusobacteria) or fungal (ascomycetes / hemiascomycetes, basidiomycetes, zygomycetes), or viral, and the occurrence of exacerbations over a period of 12 months.

DETAILED DESCRIPTION:
Therapeutic advances and the organization of care within the "CRCM" have led to an overall improvement in the management of cystic fibrosis. The protein therapies that have marked this progression only target certain genes and concern a small number of patients. The morbidity, mortality and social cost of cystic fibrosis are still considerable. Exacerbations modulate the prognosis of the disease.

We are interested in dysbiosis, which is the association of an imbalance in the composition and functions of commensal complex microbial communities and an alteration of the immune response of the host. It is involved in the development of chronic pulmonary pathologies such as cystic fibrosis Pulmonary microbiota and host responses mutually influence each other, and evidence suggests that changes in microbiota-host interactions play a major role in the evolution of chronic respiratory diseases. The response of the host may be partially measured by protein markers of inflammation or metabolites regulating inflammation (tryptophan metabolites).

Most microbiome studies focus on the bacterial microbiota, while other microorganisms such as fungi and viruses represent an important cofactor in the degradation of respiratory function. Viral dysbiosis probably plays a role in the appearance of exacerbation.

Among the few studies incorporating fungal risk, very few have considered the role of Pneumocystis jirovecii (PCJ). This non-culturable species was found in 12.5% of patients with cystic fibrosis and possibly associated with exacerbations. We will prospectively follow a cohort of cystic fibrosis patients by collecting clinical and microbiological data on various samples (exhaled air condensate (EAC), sputum and serum) on a quarterly basis and during episodes of exacerbations.

Our project will verify the hypothesis of a correlation between the microbiota, inflammation, and the production of metabolites regulating inflammation (dysbiosis), but also to determine what is the initial biological process leading to the exacerbation: dysbiosis induced by variation of the microbiota or dysbiosis induced by modification of host defense systems. In addition, unlike studies in this area, we will be interested in the bacterial, viral and fungal microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cystic fibrosis
* Patient agreeing to participate in the study
* Patient with at least 2 exacerbations in the year prior to inclusion (2 antimicrobial treatments at home or in hospital during the last 12 months)
* Patient or legal guardian of the patient able to read and understand the procedure and able to express his / her consent for the study protocol
* Stable patients, away from exacerbation (at 4 weeks from the beginning of exacerbation, found to be resolved by the investigator)
* Patient affiliated to the social security scheme

Exclusion Criteria:

* Patients who can not read
* Patients opposing the use of their medical data
* Unstable patients, less than one month from the beginning of the exacerbation
* Pregnant or lactating women
* Adult patient under curatorship or tutorship, person deprived of liberty
* Patient awaiting transplant or non-invasive ventilation in chronic
* Patient can not be contacted in case of emergency

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients followed for cystic fibrosis are followed in "CRCM". The selection of patients will be done by the various investigating physicians during consultations, day hospitals or admission to the hospital for differents reasons. This research protocol fits as much as possible in the context of routine care, particularly with respect to the rhythmicity of the various visits
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-10-02 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Identification of markers of bacterial fungal and viral dysbiosis associated with the occurrence of exacerbation in patients followed for cystic fibrosis. | One year
  Association between a modification of at least 10% of the relative abundance of a bacterial phylum (Proteobacteria, Firmicutes, Actinobacteria, Bacteroidetes, Fusobacteria) or fungal (ascomycetes / hemiascomycetes, basidiomycetes, zygomycetes), or viral and the occurrence of exacerbations over a period of 12 months.

SECONDARY OUTCOMES:
Evaluation of the influence of the modification of the relative abundance of different bacterial, viral and fungal taxa, on the occurrence of exacerbations | One year
  Association between a change of at least 10% in the relative abundance of a bacterial or fungal taxum, and the occurrence of exacerbations over a 12-month period
Evaluation of the influence of the global biodiversity of the bacterial and fungal pulmonary microbiome on the occurrence of exacerbations. | One year
  Association between a modification of two indices (Faith's Phylogenetic Diversity and Shannon's B H index) and the occurrence of exacerbations over a 12-month period
Association between markers of respiratory function and the relative abundance of different bacterial, viral and fungal phyla and taxa | One year
  Correlation between FEV1 on the one hand, and changes in the relative abundance of bacterial, viral and fungal phyla and taxa on the other hand
Evaluation of the link between an increase in inflammatory markers and the occurrence of exacerbations | One year
  Association between serum concentrations of serum inflammatory cytokines and the occurrence of exacerbations over a period of 12 months
Association between markers of respiratory function and serum inflammatory markers | One year
  Correlation between FEV 1 and CV on the one hand, and different serum inflammatory serum cytokines
Comparison of two types of sputum samples versus expired air condensate to evaluate the pulmonary microbiome in patients with cystic fibrosis | One year
  Comparison of relative abundance of phyla of interest in sputum vs exhaled air condensate
Evaluation of the interactions between the different taxa of the pulmonary microbiome of patients with cystic fibrosis | One year
  Network co-occurrence (network interference) of the relative abundance of different bacterial and fungal taxa
Evaluation of the impact of treatments administered during exacerbations on the pulmonary microbiome, in particular on changes in the relative abundance and diversity of different bacterial, viral and fungal taxa | One year
  Comparison of the relative abundance of the phyla of interest and the diversity of the microbiome (Faith's Phylogenetic Diversity and Shannon B H index) in the presence or absence of antimicrobial and anti-inflammatory steroid treatments

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beaumier L, Chanoine S, Camara B, Pison C, Bedouch P. Alemtuzumab and de novo pulmonary arterial hypertension: A potential association? J Heart Lung Transplant. 2017 Mar;36(3):370-371. doi: 10.1016/j.healun.2016.10.013. Epub 2016 Oct 29. No abstract available. PMID 27889369
- [Background] Wintenberger C, Maubon D, Charpentier E, Rendu J, Pavese P, Augier C, Malvezzi P, Camara B, Mallaret MR, Bouillet L, Epaulard O. Grouped Cases of Pulmonary Pneumocystosis After Solid Organ Transplantation: Advantages of Coordination by an Infectious Diseases Unit for Overall Management and Epidemiological Monitoring. Infect Control Hosp Epidemiol. 2017 Feb;38(2):179-185. doi: 10.1017/ice.2016.274. Epub 2016 Nov 28. PMID 27890037
- [Background] Zhao Y, Garnaud C, Brenier-Pinchart MP, Thiebaut-Bertrand A, Saint-Raymond C, Camara B, Hamidfar R, Cognet O, Maubon D, Cornet M, Perlin DS. Direct Molecular Diagnosis of Aspergillosis and CYP51A Profiling from Respiratory Samples of French Patients. Front Microbiol. 2016 Jul 29;7:1164. doi: 10.3389/fmicb.2016.01164. eCollection 2016. PMID 27524978
- [Background] Decorte N, Gruet M, Camara B, Quetant S, Mely L, Vallier JM, Verges S, Wuyam B. Absence of calf muscle metabolism alterations in active cystic fibrosis adults with mild to moderate lung disease. J Cyst Fibros. 2017 Jan;16(1):98-106. doi: 10.1016/j.jcf.2016.05.010. Epub 2016 Jun 15. PMID 27316662
- [Background] Claustre J, Brion JP, Quetant S, Bedouch P, Pison C, Camara B. Favorable Evolution of Cryptococcal Meningitis in the Context of Flucytosine Resistance. Exp Clin Transplant. 2018 Feb;16(1):110-113. doi: 10.6002/ect.2015.0217. Epub 2016 Apr 26. PMID 27143150
- [Background] Roca A, Oluwalana C, Bojang A, Camara B, Kampmann B, Bailey R, Demba A, Bottomley C, D'Alessandro U. Oral azithromycin given during labour decreases bacterial carriage in the mothers and their offspring: a double-blind randomized trial. Clin Microbiol Infect. 2016 Jun;22(6):565.e1-9. doi: 10.1016/j.cmi.2016.03.005. Epub 2016 Mar 26. PMID 27026482
- [Background] Godet C, Laurent F, Bergeron A, Ingrand P, Beigelman-Aubry C, Camara B, Cottin V, Germaud P, Philippe B, Pison C, Toper C, Carette MF, Frat JP, Beraud G, Roblot F, Cadranel J; ACHROSCAN Study Group. CT Imaging Assessment of Response to Treatment in Chronic Pulmonary Aspergillosis. Chest. 2016 Jul;150(1):139-47. doi: 10.1016/j.chest.2016.02.640. Epub 2016 Feb 19. PMID 26905365
- [Background] Dumollard C, Bailly S, Perriot S, Brenier-Pinchart MP, Saint-Raymond C, Camara B, Gangneux JP, Persat F, Valot S, Grenouillet F, Pelloux H, Pinel C, Cornet M. Prospective Evaluation of a New Aspergillus IgG Enzyme Immunoassay Kit for Diagnosis of Chronic and Allergic Pulmonary Aspergillosis. J Clin Microbiol. 2016 May;54(5):1236-42. doi: 10.1128/JCM.03261-15. Epub 2016 Feb 17. PMID 26888904
- [Background] Godet C, Laurent F, Beraud G, Toper C, Camara B, Philippe B, Germaud P, Cottin V, Beigelman-Aubry C, Khalil A, Blouin P, Pouriel M, Roblot F, Bergeron A, Cadranel J; ACHROSCAN study group. Phenotyping chronic pulmonary aspergillosis by cluster analysis. Eur Respir J. 2015 Nov;46(5):1509-12. doi: 10.1183/13993003.00869-2015. Epub 2015 Sep 17. No abstract available. PMID 26381520
- [Background] Gruet M, Decorte N, Mely L, Vallier JM, Camara B, Quetant S, Wuyam B, Verges S. Skeletal muscle contractility and fatigability in adults with cystic fibrosis. J Cyst Fibros. 2016 Jan;15(1):e1-8. doi: 10.1016/j.jcf.2015.05.004. Epub 2015 May 29. PMID 26033387
- [Background] Bouvaist H, Thony F, Jondot M, Camara B, Jais X, Pison C. Balloon pulmonary angioplasty in a patient with chronic thromboembolic pulmonary hypertension. Eur Respir Rev. 2014 Sep;23(133):393-5. doi: 10.1183/09059180.00000514. No abstract available. PMID 25176976
- [Background] Claustre J, Quetant S, Camara B, France M, Schummer G, Bedouch P, Pavese P, Saint Raymond C, Bardy B, Masson D, Roth H, Pison C; Grenoble Lung Transplantation group. Nonspecific immunoglobulin replacement in lung transplantation recipients with hypogammaglobulinemia: a cohort study taking into account propensity score and immortal time bias. Transplantation. 2015 Feb;99(2):444-50. doi: 10.1097/TP.0000000000000339. PMID 25099705
- [Background] Bosc C, Clement M, Deroux A, Mammar A, Pison C, Camara B. [Severe pneumonia due to cytomegalovirus in chronic obstructive pulmonary disease]. Rev Mal Respir. 2014 May;31(5):435-8. doi: 10.1016/j.rmr.2013.09.013. Epub 2013 Dec 2. French. PMID 24878160
- [Background] Camara B, Reymond E, Saint-Raymond C, Roth H, Brenier-Pinchart MP, Pinel C, Cadranel J, Ferretti G, Pelloux H, Pison C; Grenoble Aspergillus Committee. Characteristics and outcomes of chronic pulmonary aspergillosis: a retrospective analysis of a tertiary hospital registry. Clin Respir J. 2015 Jan;9(1):65-73. doi: 10.1111/crj.12105. Epub 2014 Feb 17. PMID 24406138